CLINICAL TRIAL: NCT06620120
Title: Single-centre, Prospective, Randomised, Controlled, Study to Investigate the Effect of EPITACT® Light Legs Therapeutic Insoles by Millet Innovation on the Symptoms and Quality of Life of Patients With Chronic Venous Disease
Brief Title: Investigate the Effect of EPITACT® Light Legs Therapeutic Insoles on the Symptoms and Quality of Life of Patients With Chronic Venous Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Millet Innovation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01923-42
Record Dates: First submitted 2024-08-22; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Venous Disease; Quality of Life; Symptoms and Signs
Keywords: chronic venous disease, insoles, quality of life, symptom, relief
MeSH Terms: conditions — Signs and Symptoms | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One medical device as investigational device (Experimental)
  Interventions: Device: Insoles
- Without device (Experimental)
  Interventions: Other: Without insoles

INTERVENTIONS:
Device: Insoles — At the D0 visit, if the patient is assigned to the arm with insoles.
  The patient completes the quality of life and symptom evaluation questionnaires, the plesthysmographic evaluation test, the analysis of walking without insoles and the oedema measurement.
  Then, at D30, the patient repeated the same tests, with the exception of the gait and plesthysmographic evaluation tests.
  The patient then switched to the other arm.
  Arms: One medical device as investigational device
Other: Without insoles — At the D0 visit, if the patient is assigned to the arm without insoles.
  The patient completes the quality of life and symptom evaluation questionnaires, the plesthysmographic evaluation test, the analysis of walking without insoles and the oedema measurement.
  Then, at D30, the patient repeated the same tests, with the exception of the gait and plesthysmographic evaluation tests.
  The patient then switched to the other arm.
  Arms: Without device

SUMMARY:
The main objective is to evaluate the effect of wearing the insoles developed by Millet Innovation on the symptoms and quality of life of patients suffering from chronic venous disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic venous disease at CEAP C2S stage - the S means that patients must be symptomatic
* Women or men aged over 18
* Good general state of health
* High or average level of activity estimated by the GAPQ questionnaire
* Patient able to understand the requirements of the trial and having signed a free and informed consent prior to study entry
* Patient able to read and understand written instructions
* Patient able to complete the self-assessment questionnaires
* Patient with a foot size between 36 and 44

Exclusion Criteria:

* Low level of activity estimated by the GAPQ questionnaire
* Cardiac, inflammatory, liver, kidney and arterial disease
* Subject with non-venous oedema
* Subject with an open wound on the foot
* Subject unable to attend all 3 visits
* Patients unable to comply with the constraints of the protocol, in particular patients whose mental state does not allow them to understand the nature, objectives and possible consequences of the study.
* Pregnant or breastfeeding women or women who are expecting to become pregnant during the study.
* Persons deprived of their liberty by a judicial or administrative decision, persons hospitalised without consent
* Adults subject to a legal protection measure or unable to express their consent
* Any other reason which, in the opinion of the investigator, could interfere with the proper conduct of the study.
* Patient unable to wear shoes with a drop of less than 2.5cm for the duration of the study
* Subject already wearing orthopaedic insoles or standard insoles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | At Day 0 then Day 30 and Day 60
  CIVIQ (ChronIc Venous Insufficiency quality of life Questionnaire) 14 : It is a quality of life assessment scale comprising 14 items grouped into four main dimensions (pain, physical, psychological, social) with 5 levels (1 point (min) to 5 points (max)).The final score is between 14 and 70 points. A low score indicates a low impact of the disease on quality of life.
Quality of life generic questionnaire | At Day 0 then Day 30 and Day 60
  The 5-level EQ-5D version (EQ-5D-5L) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1 point), to extreme problems (5 points). A low score indicates a low impact of the disease on quality of life.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' (100/100) and 'The worst health you can image' (0/100).

SECONDARY OUTCOMES:
Symptoms evaluation questionnaire | At Day 0 then Day 30 and Day 60
  Veines-sym (VEinous INsefficency Epidemologic and Economic Study - Symptoms). 26-item Anglo-Saxon scale to explore symptoms, limitations in daily activities (physical and social dimensions) and the psychological impact of CVD. The final score is between 0 and 50 points. Higher values indicate better results.
Assessment of the 'ejection fraction' of the venous blood volume (ml) | At Day 0 then Day 30 and Day 60
  Strain-gauge plethysmography around the ankle.
Leg Oedema evaluation | At Day 0 then Day 30 and Day 60
  Assessment of leg oedema by a simple and reproducible method of assessing calf volume (cm3), which is calculated from the circumferential measurements of the ankles and calves and the height between the first and last circumference taken using a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Beliard, Medical doctor, Principal Investigator — Centre Hospitalier Louis Pasteur 39100 Dole
Locations (1):
- Centre Hospitalier Louis Pasteur, Dole, France